CLINICAL TRIAL: NCT00442390
Title: Effects of Cortisol on Carbohydrate, Lipid, and Protein Metabolism; Studies of Acute Cortisol Withdrawal in Adrenocortical Failure.
Brief Title: Metabolic Effects of Acute Cortisol Withdrawal in Adrenal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1998/4375
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Addison Syndrome
Keywords: Cortisol; adrenal insufficiency; glucose metabolism; protein metabolism; lipid metabolism; insulin sensitivity.
MeSH Terms: conditions — Adrenal Insufficiency; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hydrocortisone substitution therapy versus withdrawal

SUMMARY:
Effects of adrenal steroids is generelly drawn from studies of hypercortisolism. The effects of physiological cortisol substitution and withdrawal is studied and related to the clinical syndrome of adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Female adrenal failure
* Age 18-50
* Written informed content

Exclusion Criteria:

* Diabetes mellitus
* Cancer
* Thromboembolic events
* Pregnancy and lactation
* Heart disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 2002-01; Study Completion 2003-01

PRIMARY OUTCOMES:
insulin sensitivity
local protein turnover
whole body protein turnover
glucose metabolism
serum metabolites
serum hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Jens Juel Christiansen, PhD, Principal Investigator — University of Aarhus; Claus H Gravholt, MD, Study Chair — University of Aarhus; Christian B Djurhuus, PhD, Study Chair — University of Aarhus; Per Iversen, PhD, Study Chair — University of Aarhus; Jens S Christiansen, Professor, Study Chair — University of Aarhus; Ole Schmidt, Professor, Study Chair — University of Aarhus; Jørgen Weeke, Professor, Study Chair — University of Aarhus; Jens OL Jørgensen, MD, Study Chair — University of Aarhus; Niels Møller, Professor, Study Director — University of Aarhus